CLINICAL TRIAL: NCT00515255
Title: Open-Label Exploratory Investigation Of NPL-2003 In Adolescents With Obsessive Compulsive Disorder
Brief Title: Study of NPL-2003 in Adolescents With Obsessive Compulsive Disorder (OCD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment Goal of 20 Not Met
Sponsor: Neuropharm (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPL-2003-1-POCD-001
Record Dates: First submitted 2007-08-10; First posted 2007-08-13 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Obsessive Compulsive Disorder; Neuropharm; NPL-2003
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Minocycline

INTERVENTIONS:
Drug: Minocycline — Capsules

SUMMARY:
The purpose of this study is to investigate the effect of NPL-2003 on the symptoms of Obsessive Compulsive Disorder (OCD) in an adolescent population.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for Obsessive Compulsive Disorder.
* CY-BOCS score of greater or equal to 16 at screening.
* NIMH Global OC Scale score of 7 or higher at screening.

Exclusion Criteria:

* Patients planning to commence cognitive behaviour therapy during the period of the study or those who have begun cognitive behaviour therapy within 8 weeks prior to enrolment.
* Autistic Disorder or Pervasive Developmental Disorder.
* Moderate or severe mental retardation.
* Severe renal insufficiency.

Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2007-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The change in OCD symptoms using CY-BOCS | Throughout the study

SECONDARY OUTCOMES:
The Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) | Throughout the study
NIMH Global OC Scale | Throughout the study
Clinical Global Impressions of Improvement (CGI-I) | Throughout the study
The Children's Depression Rating Scale (CDRS-R) | Throughout the study
Columbia Suicide-Severity Rating Scale (SSRS) | Throughout the study
Multidimensional Anxiety Scale for Children (MASC) | Throughout the study
Global Assessment Scale for Children (CGAS) | Throughout the study

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - New York State Psychiatric Institute, Columbia University, New York, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio